CLINICAL TRIAL: NCT06736873
Title: Effect of Light Color on Stress, Anxiety, and Psychological Well-being During Nonstress Test in Pregnant Women at Risk: A Randomized Placebo-controlled Study
Brief Title: Effect of Light Color on Stress, Anxiety, and Psychological Well-being During Nonstress Test in Pregnant Women at Risk
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Osmaniye Korkut Ata University (Other)
Responsible Party: Principal Investigator, Emine Yıldırım, Assistant professor, Osmaniye Korkut Ata University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 205323
Record Dates: First submitted 2024-12-05; First posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Pregnant Women; Stress; Light

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- light application (Experimental): Non-stress test was performed under 100 lx light application.
  Interventions: Other: Light intervention
- control group (Placebo Comparator): Non-stress test was performed under 440 lx light application.
  Interventions: Other: Light intervention

INTERVENTIONS:
Other: Light intervention — Light intervention

SUMMARY:
Purpose of the research:

To determine the effect of light color on stress, anxiety, and psychological well-being during the Nonstress Test in at-risk pregnant women. This research was planned as a single-blind randomized controlled experimental type study by comparing separate groups in the form of experiment-placebo control. Data will be collected with the Introductory Information Form, Psychological Well-being Scale, Perceived Stress Scale (PSS/PSS-14), State Trait Anxiety Inventory (STAI). The NST device is used to follow up pregnant women in the last 3 months of pregnancy, first monthly, then every two weeks and once a week. In other words, the procedure is routinely performed on every pregnant woman who comes for control. It is a device that shows the well-being of the baby and whether the mother has contractions. It is attached to the pregnant woman's abdominal area and does not cause any harm. It is not an invasive procedure. Pregnant women in the last 3 months of pregnancy who come to have NST for follow-up will be randomly selected and divided into 2 groups. A lamp with adjustable light level with Unit Unit Ut-383 Mini Luxmeter (Light Meter) will be placed in the intervention and control groups and the light level of the lamp will be adjusted to 100 lux. NST will be taken under cold (bluish white) light for the control group and under medium warm white (daylight white) light for the intervention group. Pre-test before the application and post-test after the application will be applied. The application is an invasive application that will not disturb the pregnant woman.

ELIGIBILITY:
Inclusion Criteria:

* Being at risk of pregnancy,
* being in the last trimester of pregnancy,
* being a volunteer.

Exclusion Criteria:

* Having any problem that prevents communication (such as not knowing Turkish, having hearing, speaking and understanding disorders),
* being on psychiatric treatment (pharmacotherapy or psychotherapy),
* having a disease in their eyes that prevents them from seeing

Ages: 18 Hours to 45 Hours | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2024-12-25 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-01-15 (Estimated)

PRIMARY OUTCOMES:
stress scale | 2 minutes
  questionnaire
anxiety scale | 2 minutes
  questionnaire
psychological well-being scale | 1 minutes
  questionnaire

IPD SHARING:
Plan to Share IPD: No
Can be shared when necessary.